CLINICAL TRIAL: NCT03764475
Title: A Phase 2, Multicenter, Open-Label Extension Study of the Long-Term Safety of ARQ-151 Cream 0.3% in Adult Subjects With Chronic Plaque Psoriasis Who Have Completed Preceding Study ARQ-151-201 Phase 2 Randomized Controlled Trial (Cohort 1) and Non-ARQ-151-201 Subjects (Cohort 2)
Brief Title: Long-Term Safety of ARQ-151 Cream in Adult Subjects With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-151-202
Record Dates: First submitted 2018-11-30; First posted 2018-12-05 (Actual); Results first posted 2022-08-18 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Roflumilast

STUDY DESIGN:
Intervention Model Description: Note: Subjects that consent to enter this open-label safety study have previously completed a companion study (ARQ-151-201 Phase 2 randomized controlled trial)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Long-term Safety of Roflumilast (Other): Participants applied roflumilast (ARQ-151) cream 0.3% once daily for 52 weeks
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast — Roflumilast cream 0.3% for topical application
  Other Names: ARQ-151

SUMMARY:
This is an open-label, long-term safety study of roflumilast (ARQ-151) 0.3% cream in subjects with chronic plaque psoriasis involving up to 25% total Body Surface Area (BSA). Study medication will be applied by the qualifying subjects topically once daily for 52 weeks at home. Periodic clinic visits will include assessments for clinical safety, application site reactions, and disease improvement or progression.

DETAILED DESCRIPTION:
Cohort 1 of this study consisted of participants who previously completed study ARQ-151-201 (NCT03638258), and Cohort 2 consisted of participants who were not previously enrolled in ARQ-151-201.

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent
2. Males and females ages 18 years and older
3. Subjects with chronic plaque psoriasis who met eligibility criteria for ARQ-151-201, successfully completed ARQ-151-201 through Week 12, and are able to enroll into this long-term safety study on the Week 12 visit of the previous study (ARQ-151-201).
4. Females of childbearing potential (FOCBP) must have a negative urine pregnancy test at all study visits. In addition, sexually active FOCBP must agree to use at least one form of highly effective contraception throughout the trial. Highly effective forms of contraception include: oral/implant/injectable/transdermal contraceptives, intrauterine device, or partner's vasectomy. If barrier methods are used (e.g., condom with spermicide, diaphragm with spermicide), then 2 forms of conception are required. The use of abstinence as a contraceptive measure is acceptable as long as this is a consistent part of a lifestyle choice and a backup method has been identified if the subject becomes sexually active.
5. Post-menopausal women with spontaneous amenorrhea for at least 12 months or have undergone surgical sterilization (permanent sterilization methods include hysterectomy, bilateral oophorectomy, hysteroscopic sterilization, bilateral tubal ligation or bilateral salpingectomy).

Exclusion Criteria:

1. Subjects who experienced an ARQ-151 treatment-related AE or a serious AE (SAE) that precluded further treatment with ARQ-151 cream in Study ARQ-151-201.
2. Subjects that use any Excluded Medications and Treatments
3. Current diagnosis of guttate, erythrodermic/exfoliative, palmoplantar, or pustular psoriasis.
4. Subjects who cannot discontinue the use of strong P-450 cytochrome inhibitors e.g., indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, saquinavir, suboxone and telithromycin during the study period.
5. Subjects who cannot discontinue the use of strong P-450 cytochrome inducers e.g., efavirenz, nevirapine, glucocorticoids, barbiturates (including phenobarbital), phenytoin, and rifampin during the study period.
6. Known or suspected:

   * severe renal insufficiency or severe hepatic disorders
   * hypersensitivity to component(s) of the investigational products
   * history of severe depression, suicidal ideation
7. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
8. Subjects with any serious medical condition or laboratory abnormality that would prevent study participation or place the subject at significant risk, as determined by the Investigator.
9. Subjects with a history of chronic alcohol or drug abuse within 6 months of initiation of study medication.
10. Current or a history of cancer within 5 years with the exception of fully treated skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix.
11. Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics
Locations (30):
- United States (20):
  - Arcutis Clinical Site 35, Beverly Hills, California
  - Arcutis Clinical Site 29, Northridge, California
  - Arcutis Clinical Site 28, San Diego, California
  - Arcutis Clinical Site 27, Santa Monica, California
  - Arcutis Clinical Site 12, Miami, Florida
  - Arcutis Clinical Site 16, Sanford, Florida
  - Arcutis Clinical Site 21, Louisville, Kentucky
  - Arcutis Clinical Site 34, Clinton Township, Michigan
  - Arcutis Clinical Site 33, Detroit, Michigan
  - Arcutis Clinical Site 20, Fridley, Minnesota
  - Arcutis Clinical Site 22, New York, New York
  - Arcutis Clinical Site 14, High Point, North Carolina
  - Arcutis Clinical Site 39, Bexley, Ohio
  - Arcutis Clinical Site 15, Pittsburgh, Pennsylvania
  - Arcutis Clinical Site 19, College Station, Texas
  - Arcutis Clinical Site 37, Houston, Texas
  - Arcutis Clinical Site 13, Houston, Texas
  - Arcutis Clinical Site 23, San Antonio, Texas
  - Arcutis Clinical Site 24, Webster, Texas
  - Arcutis Clinical Site 31, Norfolk, Virginia
- Canada (10):
  - Arcutis Clinical Site 18, Surrey, British Columbia
  - Arcutis Clinical Site 11, Surrey, British Columbia
  - Arcutis Clinical Site 38, Winnipeg, Manitoba
  - Arcutis Clinical Site 10, Ajax, Ontario
  - Arcutis Clinical Site 25, London, Ontario
  - Arcutis Clinical Site 26, Markham, Ontario
  - Arcutis Clinical Site 32, Oakville, Ontario
  - Arcutis Clinical Site 17, Peterborough, Ontario
  - Arcutis Clinical Site 30, Waterloo, Ontario
  - Arcutis Clinical Site 36, Windsor, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 30 study sites in the United States and Canada.
Groups:
- Cohort 1: Study 201 Participants: This arm consisted of participants who previously participated in Study ARQ-151-201 and received either roflumilast (ARQ-151) cream (0.15% or 0.3%) or vehicle cream, and agreed to enroll in the 202 study. Upon completing the 201 study, participants applied roflumilast cream 0.3% once daily for 52 weeks for long-term safety monitoring in the 202 study.
- Cohort 2: Non-study 201 Participants: This arm consisted of participants who did not previously participate in Study ARQ-151-201, and were enrolled in the 202 study after the time of amendment 1. Participants applied roflumilast cream 0.3% once daily for 52 weeks for long-term safety monitoring.
Period: Overall Study
Arm/Group | Cohort 1: Study 201 Participants | Cohort 2: Non-study 201 Participants
Started | 230 | 102
Completed | 164 | 80
Not Completed | 66 | 22
Not completed — Adverse Event | 11 | 2
Not completed — Lost to Follow-up | 24 | 10
Not completed — Withdrawal by Subject | 26 | 10
Not completed — Lack of Efficacy | 3 | 0
Not completed — COVID-19 Disruption | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline was defined as the last observation prior to administration of ARQ-151 cream. Thus the baseline assessments for participants in Cohort 1 assigned to ARQ-151 cream occurred in the ARQ-151-201 study, whereas baseline occurred in this study (ARQ-151-202) for vehicle cream participants in the 201 study and Cohort 2 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Study 201 Participants | Cohort 2: Non-study 201 Participants | Total
Number analyzed (Participants) | 230 | 102 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (13.52) | 52.7 (15.64) | 54.5 (14.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 46 | 150
  Male | 126 | 56 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 17 | 63
  Not Hispanic or Latino | 184 | 84 | 268
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 6 | 19
  Black or African American | 24 | 5 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 183 | 85 | 268
  Multiple/Other | 10 | 5 | 15
Modified Psoriasis Area Severity Index (mPASI) [Mean (Standard Deviation); unit: score on a scale] — The mPASI combines the assessment of the severity of lesions and the area affected into a single score ranging from 0 ('no disease') to 72 ('maximal disease'), with higher scores indicating greater severity. Population: One participant in Cohort 2 did not have a baseline mPASI assessment.
  score on a scale
    number analyzed (Participants) | 230 | 101 | 331
    (all) | 5.42 (3.700) | 4.50 (3.821) | 5.14 (3.755)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing ≥1 Treatment-emergent Adverse Event (TEAE)
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. All AEs that began after initiating study treatment (treatment-emergent AEs [TEAEs]) in ARQ-151-202 are presented.
Time Frame: Up to 52 weeks
Population: All randomized participants who received ≥1 dose of study treatment are included.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Non-study 201 Participants: This arm consisted of participants who did not previously participate in study ARQ-151-201, and were enrolled after the time of amendment 1 in this study. Participants applied roflumilast cream 0.3% once daily for 52 weeks to monitor long-term safety.
Arm/Group | Cohort 1: Study 201 Participants | Cohort 2: Non-study 201 Participants
Number analyzed (Participants) | 230 | 102
Participants | 104 | 60

2. Primary Outcome: Number of Participants Experiencing ≥1 Serious Adverse Event (SAE)
Description: An SAE is any AE that in the view of either the PI or Sponsor, results in any of the following outcomes: Death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Up to 52 weeks
Population: All randomized participants who received ≥1 dose of study drug are included.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Study 201 Participants: This arm consisted of participants who previously participated in study ARQ-151-201 and received either ARQ-151 cream (0.15% or 0.3%) or vehicle cream, and agreed to enroll in the 202 study. Upon completing the 201 study, participants applied ARQ-151 cream 0.3% once daily for 52 weeks for long-term safety monitoring in the 202 study.
- Cohort 2: Non-study 201 Participants: This arm consisted of participants who did not previously participate in study ARQ-151-201, and were enrolled in the 202 study after the time of amendment 1. Participants applied ARQ-151 cream 0.3% once daily for 52 weeks for long-term safety monitoring.
Arm/Group | Cohort 1: Study 201 Participants | Cohort 2: Non-study 201 Participants
Number analyzed (Participants) | 230 | 102
Participants | 8 | 2

3. Secondary Outcome: Number of Participants With an Investigator Global Assessment (IGA) Score of 'Clear' or 'Almost Clear'
Description: The number of participants with an IGA score of 0 ('clear') or 1 ('almost clear') at Week 12 is reported. The IGA is a 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater plaque severity.
Time Frame: Weeks 12, 24, 36, and 52
Population: All participants who received ≥1 dose of study drug and have data available at the relevant time points are included.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Study 201 Participants: This arm consisted of participants who previously participated in study ARQ-151-201 and received either roflumilast cream (0.15% or 0.3%) or vehicle cream, and agreed to enroll in the 202 study. Upon completing the 201 study, participants applied roflumilast cream 0.3% once daily for 52 weeks for long-term safety monitoring in the 202 study.
Arm/Group | Cohort 1: Study 201 Participants | Cohort 2: Non-study 201 Participants
Number analyzed (Participants) | 209 | 95
Participants
  Week 12 | 92 | 47
  Week 24: number analyzed (Participants) | 189 | 87
  Week 24 | 79 | 34
  Week 36: number analyzed (Participants) | 178 | 79
  Week 36 | 68 | 36
  Week 52: number analyzed (Participants) | 165 | 81
  Week 52 | 68 | 39

4. Secondary Outcome: Duration of Response in Participants Achieving 'Clear' IGA Score
Description: The median time to re-starting study therapy among participants who achieve a 'clear' IGA score and stop treatment to all lesions is presented.
Time Frame: Up to 52 weeks
Population: All participants who received ≥1 dose of study drug and achieved an IGA score of 'clear' are included.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 1: Study 201 Participants | Cohort 2: Non-study 201 Participants
Number analyzed (Participants) | 23 | 6
weeks | 8.0 [4.1 to 9.0] | 12.4 [3.0 to NA] — Upper bound of the 95% CI was not estimable due to low number of cases.

5. Secondary Outcome: Number of Participants With Intertriginous Area Involvement Achieving an Intertriginous Area Investigator Global Assessment (I-IGA) Score of "Clear' or 'Almost Clear'
Description: The number of participants who had intertriginous area involvement with an I-IGA score of 'clear' or 'almost clear' is presented. The I-IGA is 5-point scale assessing the severity of plaque psoriasis in the intertriginous area, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater plaque severity.
Time Frame: Weeks 12, 24, 36, and 52
Population: All participants who received ≥1 dose of study drug, have intertriginous area involvement, and have data available at the relevant time points are included. This endpoint was added at protocol amendment 1, and thus I-IGA was not assessed in a subset of participants in Cohort 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Study 201 Participants | Cohort 2: Non-study 201 Participants
Number analyzed (Participants) | 38 | 26
Participants
  Week 12: number analyzed (Participants) | 16 | 25
  Week 12 | 11 | 15
  Week 24: number analyzed (Participants) | 33 | 26
  Week 24 | 13 | 14
  Week 36: number analyzed (Participants) | 38 | 20
  Week 36 | 13 | 10
  Week 52: number analyzed (Participants) | 37 | 21
  Week 52 | 9 | 10

6. Secondary Outcome: Number of Participants Achieving a 75% Reduction From Baseline in Modified Psoriasis Severity Index (mPASI-75)
Description: The number of participants achieving a 75% reduction in mPASI (eg, mPASI-75) score relative to baseline is presented. The mPASI combines the assessment of the severity of lesions and the area affected into a single score ranging from 0 ('no disease') to 72 ('maximal disease'), with higher scores indicating greater severity.
Time Frame: Baseline and Weeks 12, 24, 36, and 52
Population: All participants who received ≥1 dose of study drug and have data available at the relevant time points are included. This endpoint was added at protocol amendment 1, and thus mPASI was not assessed in a subset of participants in Cohort 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Study 201 Participants | Cohort 2: Non-study 201 Participants
Number analyzed (Participants) | 230 | 102
Participants
  Week 12: number analyzed (Participants) | 91 | 95
  Week 12 | 67 | 63
  Week 24: number analyzed (Participants) | 153 | 87
  Week 24 | 114 | 57
  Week 36: number analyzed (Participants) | 178 | 79
  Week 36 | 130 | 55
  Week 52: number analyzed (Participants) | 165 | 81
  Week 52 | 124 | 61

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: All participants who received ≥1 dose of study drug are included.
Arm/Group | Cohort 1: Study 201 Participants | Cohort 2: Non-study 201 Participants
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/102
Serious Adverse Events (participants affected / at risk) | 8/230 | 2/102
Other Adverse Events (participants affected / at risk) | 15/230 | 7/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Study 201 Participants (N=230) | Cohort 2: Non-study 201 Participants (N=102)
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Device failure (Product Issues) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Study 201 Participants (N=230) | Cohort 2: Non-study 201 Participants (N=102)
Upper respiratory tract infection (Infections and infestations) | 15 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT03764475/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT03764475/SAP_001.pdf